CLINICAL TRIAL: NCT07109466
Title: Targeting the Hip Abductors to Reduce Falls in Older Veterans Through A Virtual Multimodal Balance Intervention
Acronym: Virtual MMBI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRD6-005-24W; I01RD000434 (Other Grant/Funding Number: Veteran Affairs Rehabilitation RDT Service)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Falls
Keywords: Fall

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MMBI + Gerofit (Experimental): Participation in a virtual multi-modality balance intervention that targets the hip abductors for 3-months followed by 9 months participation in virtual Gerofit
  Interventions: Other: Mulit-modality Balance Intervention; Other: Gerofit
- Gerofit (Active Comparator): Participation in a virtual wellness program that consists of a warm up, aerobic training, and general strength training
  Interventions: Other: Gerofit

INTERVENTIONS:
Other: Mulit-modality Balance Intervention — Participants will attend a virtual group balance class that focuses on movement and obstacle negotiation 3 times per week for 3-months
  Other Names: MMI
  Arms: MMBI + Gerofit
Other: Gerofit — Participation in a virtual wellness program that consists of a warm up, aerobic training, and general strength training 3-times per week for up to 12 months

SUMMARY:
Falls are a major health concern and a leading cause of injurious death and non-fatal injuries in older Veterans who are at greater risk for falls than non-Veterans. This in-person exercise intervention targeting changes in the hip muscles, known to play a major role in balance, has been effective at reducing falls in older Veterans. Gerofit is a VA best practice health promotion program that demonstrates good success in engaging Veterans in exercise. However, the role of Gerofit in fall prevention is unknown. Some Veterans may require additional training prior to participation in Gerofit to maximize the benefits of Gerofit. The proposed intervention will use novel home-based methods of exercise to improve hip muscles prior to participating in Gerofit. The goal of this study is to evaluate if a live virtual home-based multimodal balance intervention done prior to Gerofit compared to Gerofit alone will have a greater benefit on fall risk reduction and improved muscle and mobility function.

DETAILED DESCRIPTION:
Falls are multifactorial in origin, with a failure to negotiate environmental hazards, muscle weakness, impaired postural control, and gait and balance deficits among the top contributors. Common between these is impaired lower extremity function, including difficulties during walking, incident slips and trips, or an inability to effectively recover after a loss of balance. The multifactorial origin of falls requires a multimodal approach to effectively reduce risk. The CDC currently includes 17 exercise interventions targeting fall reduction, and most of these programs reportedly decrease fall risk by ~30%. The investigators' MMBI program, developed over the last ten years, is unique in its approach to exercise for fall prevention. It has been developed in older Veterans at high risk for falls, who suffer an average of 16 comorbid health conditions. Further, the target of the hip abductors and multiple planes of movement with functional exercises and progressive lower extremity strengthening is unique to the MMBI program. While some programs have been widely studied, the majority do not have validated benefit to mechanistic outcomes, such as changes in muscle quality or intermuscular adipose tissue. In an on-going systematic review of studies that utilize a live-virtual format for fall prevention, the investigators found only 4 of 16 studies looked at falls at baseline and post-intervention. No studies utilizing the live virtual format followed individuals for a year after intervention to assess the long-term intervention effects. Most falls occur during walking, after incident slips and trips, such that targeted interventions to avoid loss of balance focused on stepping, obstacle negotiation, and walking ability -while also strengthening the muscles critical for balance recovery- are critical to reducing falls. Recent guidelines also suggest that any older adults with impaired gait or balance (slow gait speed or high TUG or FSST time) should be offered tailored exercise focused on balance, gait and strength to prevent future falls. This MMBI program is unique in that it targets not only strengthening but also functional movements in multiple plans to target the hip abductors, improve balance and reduce falls.

This study will address several important knowledge gaps, first by simply assessing the effect of the live virtual Gerofit program on balance and falls. It will also determine whether proven methods of improving balance and hip abductor strength can be safely and effectively translated to novel home delivery for Veterans, using an established standard of care control, and clinically important outcomes of fall rate, muscle strength, and muscle quality via CT scan. This will provide critical information for future fall prevention studies in the VA. In prior studies examining the effects of resistance training on balance, less than 30% of all trials included any resistance training of the hip abductors. Further, the investigators are unaware of any trial that currently targets the hip abductors with a virtual or home-based fall risk reduction intervention in a group that are at increased risk for falls. Understanding mechanistic contributions of the hip abductors to balance and mobility, and finding targeted means to improve their function without the need for center-based exercise opens important new treatment options for older Veterans with mobility limitations at increased fall risk. The investigators will do this through the following Aims.

Aim 1: Determine the 12-week effects of vMMBI vs vGerofit alone on clinical measures of fall risk, physical function, and fear of falling. It is hypothesized greater improvements in fall risk (four-square step test [primary outcome]) following 12 weeks of vMMBI compared to 12 weeks of vGerofit.

Aim 2: Determine the 12-week effects of vMMBI vs vGerofit alone on hip abductor mechanisms of fall prevention, including hip abductor function, hypertrophy, and quality. It is hypothesized that Veterans in the vMMBI group will demonstrate greater improvements in hip abductor (gluteus minimus/medius) function (muscle strength - determined with hand-held dynamometer [primary outcome]) due to the synergistic effects of resistance training combined with balance and mobility exercises, which may enhance muscle hypertrophy of the hip abductors (cross-sectional area) and improve muscle quality (% intramuscular fat by computed tomography).

Clinical Translational Aim: Determine the efficacy of participation in vMMBI+vGerofit vs vGerofit alone as indicated by the incidence of falls and exercise adherence.

ELIGIBILITY:
Inclusion Criteria:

* Veteran Status
* 65 years or older
* VA primary Care provider
* Enrolled in the VA Maryland Health Care System for health care
* At risk for Falls

Exclusion Criteria:

* Poorly controlled hypertension
* Home oxygen use
* Contraindications to exercise or resistance exercise
* Significant cognitive impairment
* Other medical condition precluding patient participation in this study as per medical judgment of study team

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-05-01 (Estimated); Study Completion 2031-05-30 (Estimated)

PRIMARY OUTCOMES:
Balance | 3-months
  The four-square step test will be used as a measure of balance. The change in the amount of time it takes to complete the four-square step test comparing pre and post-intervention.
Isometric Hip Abductor Strength | 3-months
  A measure of the maximal isometric muscle strength produced in hip abductor muscles will be assessed with a handheld dynamometer device. Pre-test levels will be compared to post-intervention levels.

SECONDARY OUTCOMES:
Mobility | 3-months
  The Timed up and Go will be used as a measure of mobility. The change in the amount of time it takes to complete the timed up and go test is comparing pre to post-intervention levels.

CONTACTS AND LOCATIONS:
Overall Officials: Odessa R. Addison, PhD DPT, Principal Investigator — Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD
Locations (1):
- Baltimore VA Medical Center VA Maryland Health Care System, Baltimore, MD, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No